CLINICAL TRIAL: NCT02120378
Title: Correlation Between Fetal Gestational Age, Viability and Survival Rates in Egypt
Brief Title: Fetal Viability Estimation in Egypt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Dina Mohamed Refaat Dakhly, MD, Cairo University
Other Study IDs: WH142014
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Premature Birth; Miscarriage
Keywords: miscarriage; fetal viability; prematurity
MeSH Terms: conditions — Premature Birth; Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Due to the discrepancy between the Egyptian and the conventional definition of miscarriage or live birth, there seemed to be a need for a study that ends up with reaching a definition for the mentioned terms. live birth is known to be for fetus born after 20 weeks or of weight more than 500 grams, while in Egypt, this is not applicable. basically the neonate has a chance of survival if the weight is more than 1000 grams or of gestational age more than 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* pregnant females age from 18- 40 years old
* preterm delivery before completing 38 weeks of gestation
* singleton or multiple gestation
* fetuses with congenital anomalies

Exclusion Criteria:

* refusal to get enrolled in the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: females presenting to the causality department in kasr el Aini hospital presenting with signs of preterm labor ( uterine contractions before completing 38 weeks of gestation)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-08 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
determination of age of fetal viability according the survival rate percentage | 1 year

SECONDARY OUTCOMES:
most common causes for premature delivery in Egypt | 6 months
the mode of delivery of preterm cases in Egypt | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: dina m dakhly, MD, Principal Investigator — Cairo University
Locations (1):
- Kasr El Aini, Cairo, Cairo Governorate, Egypt